CLINICAL TRIAL: NCT03247296
Title: Study of the Early Occurrence of Hepatocellular Carcinoma (HCC) in Egyptian HCV Infected Patients Receiving Sofosbuvir and Daclatasvir
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Aya Mohammed Mohammed Essawy, Assistant Lecturer, MTI University
Other Study IDs: 3132010
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C
Keywords: Daclatasvir; HCC; HCV; Sofosbuvir
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; daclatasvir; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Patients taking Sofosbuvir and Daclatasvir
  Interventions: Drug: Sofosbuvir 400 mg, Daclatasvir, Ribavirin
- Group B: Patients taking Sofosbuvir,Daclatasvir, and Ribavirin
  Interventions: Drug: Sofosbuvir 400 mg, Daclatasvir, Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir 400 mg, Daclatasvir, Ribavirin — No intervention made this is an observational study to monitor the already existing protocols of the facility

SUMMARY:
To evaluate the early detection of HCC in patients Taking Sofosbuvir and Daclatasvir.

DETAILED DESCRIPTION:
Methodology:

Design:

Prospective, randomized study used to detect early incidence of HCC in patients taking Sofosbuvir and Daclatasvir to treat HCV.

Patients will be recruited from the National Hepatology and Tropical Medicine Research Institute (NHTMRI)

Duration of study:

24 weeks from starting the DAAs

Methods:

Patients will go through examination and lab. Workup three times in this study:

* FIRST time:

  * Before starting antiviral therapy, all included patients will undergo through physical examination, lab workup including HCV-RNA quantitative, fasting plasma glucose or HbA1C if diabetic, serum creatinine, CBC, AST, ALT, prothrombin Concentration or INR, total bilirubin, serum albumin, Pregnancy test ( Ladies in child bearing period), AFP as a marker of HCC.
  * Included patients will also undergo through diagnostic procedures as Abdominal ultrasonography and ECG (men >40, women>50).
* Second time:

  * At the end of antiviral therapy (12 weeks), virological response to therapy will be assessed by quantitative HCV RNA detection, using PCR.
  * Patients will lab workup including , fasting plasma glucose or HbA1C if diabetic, serum creatinine, CBC, AST, ALT, prothrombin Concentration or INR, total bilirubin, serum albumin, AFP as a marker of HCC.
  * The abdominal ultrasonography will be repeated any suspected focal lesion of the liver will be evaluated with triphasic CT scan or MRI to assess the occurrence or the recurrence of HCC.
* Third and last time:

  * At 24 weeks ( Patients will be off treatment for the previous 12 weeks) , virological response to therapy will be assessed by quantitative HCV RNA detection, using PCR.
  * Patients will lab workup including, fasting plasma glucose or HbA1C if diabetic, serum creatinine, CBC, AST, ALT, prothrombin Concentration or INR, total bilirubin, serum albumin, AFP as a marker of HCC.
  * The abdominal ultrasonography will be repeated any suspected focal lesion of the liver will be evaluated with triphasic CT scan or MRI to assess the occurrence or the recurrence of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Patients have positive HCV-RNA and taking DAAS to treat it.
* Both sexes will be included
* Age above 18 to 75 years old
* Child Pugh score ( A and B )

Exclusion Criteria:

* Total serum bilirubin<3 mg/dl
* Serum albumin > 2.8 g/dl
* INR≥ 1.7
* Platelet count< 50000/mm3 IF any of the above criteria is not caused by liver disease, the patient can be included in the study.
* HCC, except 4 weeks after intervention aiming at cure with no evidence of activity by dynamic imaging (CT or MRI).
* Extra- hepatic malignancy.
* Pregnancy or inability to use effective contraception.
* Inadequately controlled diabetes mellitus (HbA1c>9%).

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients have positive HCV-RNA and taking DAAS to treat it.
  * Both sexes will be included
  * Age above 18 to 75 years old
  * Child Pugh score (A and B)
  Patients randomly enrolled in the study from the hepatitis clinic in the National Hepatology and Tropical Medicine research Institute
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-10-31 (Estimated); Study Completion 2017-11-10 (Estimated)

PRIMARY OUTCOMES:
HCC | 24 weeks
  occurence of HCC

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A Sabri, Professor, Study Chair — Professor and Head of Clinical Pharmacy Department Faculty of Pharmacy Ain Shams University; Abd El Rahman El Naggar, Professor, Study Director — Professor of clinicalpharmacology and Toxicology and Head of clinical pharmacy Department MTI University; Hasan A El Garem, Professor, Study Director — Prof. Dr. of Endemic Medicine, hepatology, and gastroenterology Faculty of Medicine Cairo University; Aya M Esawy, Assistant Lecturer, Principal Investigator — Assistant Lecturer of clinical pharmacy at faculty of pharmacy MTI university; Sara M Zaki, Lecturer, Study Director — Lecturer of clinical Pharmacy Faculty of pharmacy Ain-Shams University; May I Mehrez, Fellow, Study Director — Fellow of Hepatology Internal Medicine Department (NHTMRI)
Locations (1):
- National Hepatology and Tropical Medicine Research Institute, Cairo, Egypt